CLINICAL TRIAL: NCT04974710
Title: Developing an US-MRI Biomarker Fusion Model for Endometriosis (DEFEND)
Brief Title: Developing an US-MRI Biomarker Fusion Model for Endometriosis
Acronym: DEFEND
Status: Completed | Type: Observational
Sponsor: Perspectum (Industry)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 20/WS/0111
Record Dates: First submitted 2021-06-11; First posted 2021-07-23 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Endometriosis; Reproductive System Disorder
Keywords: Reproductive health; Diagnostics; Magnetic Resonance Imaging; Ultrasound; Biomarkers
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Outpatient MRI — All participants will undergo a standardised imaging protocol in a MRI scanner. This will take place during the same visit or following the transvaginal ultrasound (TVUS) and in advance of any surgical procedure (laparoscopy).

SUMMARY:
Single centre, prospective, observational, cohort study looking to develop a database representing the variability of disease and imaging seen in women with clinically diagnosed endometriosis, awaiting laparoscopic surgery.

DETAILED DESCRIPTION:
In the United Kingdom (UK), endometriosis is one of the most common gynaecological diseases needing treatment. The prevalence of disease is often underestimated, however it is believed to affect at least 1 in 10 women in the UK. Within the NHS, endometriosis costs the UK economy approximately £8.2 billion a year in treatment, loss of work and healthcare costs.

Currently, the first diagnostic recommendation for endometriosis is and Ultrasound (US) scan or a MRI, followed by a diagnostic surgery called laparoscopy. Accurate diagnoses is usually limited to specialist tertiary centres, therefore a delayed diagnosis is a significant problem for women with endometriosis. Limited experience in the disease area can also lead to misdiagnosis and the latest report from the National Institute of Clinical Excellence (NICE) reports a time delay of around 7.5 years before a confirmed diagnosis of endometriosis. A model that could accurately predict surgical findings of endometriosis would be of significant clinical and economical benefit.

The main aim of this study is to curate a database of patients with varying levels of endometriosis. This database will contain fully anonymised MR and US images alongside clinical data for further use in research. There will be no intervention outside of standard of care. US and clinical data will be collected during routine visits and patients will be offered an additional visit to have a MRI. The ultimate aim is to then use this data to develop a widely available diagnostic tool based on MRI and US imaging modalities using computer modelling. Validating the predictive model with surgical findings will increase confidence and access to advanced imaging for non-experts, allowing clinicians to accurately predict surgical findings as well as reduce time to diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18-40 years
* Clinically diagnosed endometriosis and awaiting surgery
* BMI 20-35 kg/m2
* No past abdominal surgical history
* Participant willing and able to give informed consent for participation in the study

Exclusion Criteria:

* Previous surgery in 12 months prior to consent:

  * abdominal surgery
  * surgery for endometriosis
* The participant may not enter the study if they have any contraindication to magnetic resonance imaging (standard MR exclusion criteria including pregnancy, extensive tattoos, pacemaker, shrapnel injury, severe claustrophobia).
* Any other cause, including a significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or may influence the participant's ability to participate in the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women with clinically diagnosed endometriosis and awaiting laparoscopic surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Build a database of 100 patients with endometriosis, awaiting confirmatory laparoscopic surgery on to an anonymised database for future use in algorithm development. | 12 months

SECONDARY OUTCOMES:
Evaluate inter-observer variability in diagnosing and staging endometriosis using both two and three dimensional ultrasound by computing inter-rater agreement statistics (e.g. Kappa statistic) | 12 months
Assess the utility multi-parametric MRI in diagnosing and staging endometriosis | 12 months
  Using measurements such as cT1, PDFF and Diffusion Weighted Imaging (DWI) to the MR imaging variables with a clinical diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Ippokratis Sarris, BM, BCh, Principal Investigator — King's Fertility
Locations (1):
- King's Fertility, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual participant will be identified.

REFERENCES:
- [Background] Bulun SE, Yilmaz BD, Sison C, Miyazaki K, Bernardi L, Liu S, Kohlmeier A, Yin P, Milad M, Wei J. Endometriosis. Endocr Rev. 2019 Aug 1;40(4):1048-1079. doi: 10.1210/er.2018-00242. PMID 30994890
- [Background] Bondza PK, Maheux R, Akoum A. Insights into endometriosis-associated endometrial dysfunctions: a review. Front Biosci (Elite Ed). 2009 Jun 1;1(2):415-28. doi: 10.2741/E38. PMID 19482656
- [Background] Johnson NP, Hummelshoj L, Adamson GD, Keckstein J, Taylor HS, Abrao MS, Bush D, Kiesel L, Tamimi R, Sharpe-Timms KL, Rombauts L, Giudice LC; World Endometriosis Society Sao Paulo Consortium. World Endometriosis Society consensus on the classification of endometriosis. Hum Reprod. 2017 Feb;32(2):315-324. doi: 10.1093/humrep/dew293. Epub 2016 Dec 5. PMID 27920089
- [Background] Heilier JF, Donnez J, Nackers F, Rousseau R, Verougstraete V, Rosenkranz K, Donnez O, Grandjean F, Lison D, Tonglet R. Environmental and host-associated risk factors in endometriosis and deep endometriotic nodules: a matched case-control study. Environ Res. 2007 Jan;103(1):121-9. doi: 10.1016/j.envres.2006.04.004. Epub 2006 Jun 15. PMID 16781705
- [Background] Koninckx PR, Martin DC. Deep endometriosis: a consequence of infiltration or retraction or possibly adenomyosis externa? Fertil Steril. 1992 Nov;58(5):924-8. doi: 10.1016/s0015-0282(16)55436-3. PMID 1426377
- [Background] Ferrero S, Alessandri F, Racca A, Leone Roberti Maggiore U. Treatment of pain associated with deep endometriosis: alternatives and evidence. Fertil Steril. 2015 Oct;104(4):771-792. doi: 10.1016/j.fertnstert.2015.08.031. Epub 2015 Sep 10. PMID 26363387
- [Background] Leyland N, Casper R, Laberge P, Singh SS; SOGC. Endometriosis: diagnosis and management. J Obstet Gynaecol Can. 2010 Jul;32(7 Suppl 2):S1-32. PMID 21545757
- [Background] Berger J, Henneman O, Rhemrev J, Smeets M, Jansen FW. MRI-Ultrasound Fusion Imaging for Diagnosis of Deep Infiltrating Endometriosis - A Critical Appraisal. Ultrasound Int Open. 2018 Sep;4(3):E85-E90. doi: 10.1055/a-0647-1575. Epub 2018 Sep 24. PMID 30255164
- [Background] Bazot M, Thomassin I, Hourani R, Cortez A, Darai E. Diagnostic accuracy of transvaginal sonography for deep pelvic endometriosis. Ultrasound Obstet Gynecol. 2004 Aug;24(2):180-5. doi: 10.1002/uog.1108. PMID 15287057
- [Background] Slack A, Child T, Lindsey I, Kennedy S, Cunningham C, Mortensen N, Koninckx P, McVeigh E. Urological and colorectal complications following surgery for rectovaginal endometriosis. BJOG. 2007 Oct;114(10):1278-82. doi: 10.1111/j.1471-0528.2007.01477.x. PMID 17877680
- [Background] Padavala J, Navaneetham N. Complications after surgery for deeply infiltrating pelvic endometriosis. BJOG. 2011 Dec;118(13):1678; author reply 1678-9. doi: 10.1111/j.1471-0528.2011.03162.x. No abstract available. PMID 22077260
- [Background] Nezhat C, Li A, Falik R, Copeland D, Razavi G, Shakib A, Mihailide C, Bamford H, DiFrancesco L, Tazuke S, Ghanouni P, Rivas H, Nezhat A, Nezhat C, Nezhat F. Bowel endometriosis: diagnosis and management. Am J Obstet Gynecol. 2018 Jun;218(6):549-562. doi: 10.1016/j.ajog.2017.09.023. Epub 2017 Oct 13. PMID 29032051
- [Background] Rosefort A, Huchon C, Estrade S, Paternostre A, Bernard JP, Fauconnier A. Is training sufficient for ultrasound operators to diagnose deep infiltrating endometriosis and bowel involvement by transvaginal ultrasound? J Gynecol Obstet Hum Reprod. 2019 Feb;48(2):109-114. doi: 10.1016/j.jogoh.2018.04.004. Epub 2018 Apr 11. PMID 29654939
- [Background] Creed JM, Maggrah A, Usher R, Desa E, Harbottle A. How can mitochondrial DNA deletions act as a biomarker for the detection of endometriosis within the clinic? Biomark Med. 2020 Jan;14(1):5-8. doi: 10.2217/bmm-2019-0435. Epub 2019 Nov 5. No abstract available. PMID 31686548
- [Background] Viera AJ, Garrett JM. Understanding interobserver agreement: the kappa statistic. Fam Med. 2005 May;37(5):360-3. PMID 15883903